CLINICAL TRIAL: NCT07375199
Title: Reducing Mental Health Stigmatization Among Healthcare Workers and Students Using a Virtual Reality Protocol: The VIRTUS Protocol, a Randomized Controlled Trial
Brief Title: Reducing Mental Health Stigmatization Among Healthcare Workers and Students Using a Virtual Reality Protocol: The VIRTUS Protocol
Acronym: VIRTUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025-A01472-47
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Disorder
Keywords: stigma; virtual reality; empathy; implicit associations
MeSH Terms: conditions — Schizophrenia; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia (Experimental): The protocol involves two short VR scenarios. In the intervention condition only ("schizophrenia"), both scenarios will simulate auditory and visual hallucinations and persecutory delusions, to immerse participants in the experience of someone living with schizophrenia.
  Interventions: Other: VIRTUS
- CONTROL (Active Comparator): The protocol involves two short VR scenarios. In the control condition participant will see the same VR video, without auditory and visual hallucinations or persecutory delusions.
  Interventions: Other: VR Control

INTERVENTIONS:
Other: VIRTUS — Participants will watch two brief VR videos. The first simulates an office environnement , the second simulates a university classroom environment. In the experimental group, psychotic-like phenomena commonly reported by individuals with schizophrenia during acute episodes (e.g., auditory hallucinations, visual hallucinations, paranoid ideation) will be incorporated into both videos. The purpose is to simulate the lived experience of schizophrenia. The two VR environnements were adapted form Marques (virtual Stroop test, Marques et al., 2022) and Abrams (University classroom, Abrams et al., 2024), and programmed using Unity2021.3.11 with C#. Some assets in scenes were developped with Blender 4.4. We used MetaQuest2 as headset VR.
  Arms: Schizophrenia
Other: VR Control — Participants will watch two brief VR videos. The first simulates an office environnement , the second simulates a university classroom environment. Contrary to the experimental group, psychotic-like phenomena (auditory hallucinations, visual hallucinations, paranoid ideation) will not be incorporated into videos. The two VR environnements are programmed using Unity2021.3.11 with C#. Some assets in scenes were developped with Blender 4.4. We used MetaQuest2 as headset VR.
  Arms: CONTROL

SUMMARY:
Schizophrenia is a chronic psychiatric disorder, frequently associated with stigma, including within healthcare settings, that significantly impairs quality of life and symptoms. Virtual Reality (VR), as an immersive tool, may allow healthy individuals to experience the first-person perspective of a patient undergoing psychotic symptoms. VR exposure may facilitate perspective-taking, fosters empathy, and studies suggest VR could be a valuable tool to reduce stigma. However, the findings remain incomplete, with considerable variation between protocols and no data on implicit stigma. This study is designed to evaluate the effectiveness of a VR protocol simulating psychotic symptoms on explicit and implicit stigma.

Methods and Analysis A randomized controlled trial involving 128 participants will be conducted. Participants will include healthcare workers and students (medicine, nursing, or psychology) recruited from CH Henri Laborit in Poitiers (France), Poitiers University Hospital, CH Nord-Deux-Sèvres in Thouars (France), and the University of Poitiers. Recruitment will take place over a two-year period. Participants will be randomly assigned to either the intervention group or the control group.

The protocol involves two short VR scenarios. In the intervention condition only, both scenarios will simulate auditory and visual hallucinations and persecutory delusions, to immerse participants in the experience of someone living with schizophrenia. Stigma will be assessed before the VR intervention, immediately afterward, and at one-month follow-up. Assessment will be conducted using self-report scales (Attribution Questionnaire-27 items by Corrigan et al., 2003 (AQ-27), Community Attitudes toward the Mentally Ill, Taylor & Dear 1981 (CAMI) and Reported and Intended Behavior Scale by Evans-Lacko et al., 2011 (RIBS) for explicit stigma, and a behavioural test (Implicit Association Task, Greenwald, McGhee et Schwartz en 1998 (IAT)) for the implicit stigma.

The primary outcome is the reduction in stigma toward individuals with schizophrenia, assessed with the AQ-27 scale, from baseline to the one-month follow-up, comparing the intervention and control groups. The expected result is a greater reduction in stigma in the intervention group compared to the control group. Secondary outcomes include a one-month reduction in implicit associations, immediate post-intervention effects on stigma, changes in self-reported prejudice and discrimination over time.

Ethics and Dissemination All participants receive both oral and written information and provided signed informed consent. The study is under review from the French Research Ethics Committee (reference number: 2025-A01472-47). Results will be disseminated through presentations, conferences, and publications in peer-reviewed scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65
* currently employed as a healthcare professional or enrolled as a advanced-grade student in medicine, nursing, or psychology
* no history of psychiatric or addictive disorders (except for tobacco dependence)
* covered by French social security
* able to provide informed written consent after receiving appropriate information.

Exclusion Criteria:

* current or past psychiatric or addictive disorder (except tobacco dependence)
* use of antipsychotic medication; first-degree family history of schizophrenia; cognitive impairment
* susceptibility to cybersickness
* recent (<1 year) or acute neurological disorders
* history of epilepsy
* known otorhinolaryngologic conditions causing vertigo, nausea or vomiting
* pregnancy or breastfeeding
* legal protection measures
* any condition, in the investigator's opinion that would prevent valid questionnaire completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Explicit stigma - 1 month follow up | Baseline and 1 month after intervention
  Change from baseline to 1 month follow-up, in the Attribution Questionnaire-27 (AQ-27) total score, comparing the intervention and control groups. Higher scores indicate greater explicit stigma toward individuals with schizophrenia.

SECONDARY OUTCOMES:
Implicit stigma - 1 month follow up | Baseline and 1 month after intervention
  Change from baseline in Implicit Association Test (IAT) score for the schizophrenia-violence association. Higher scores indicate a stronger implicit association in the direction defined by the scoring algorithm.
  A greater reduction in implicit associations, as measured by the IAT, is expected at one month in the intervention group compared with the control group.
Explicit stigma - Immediate effect | Baseline (pre-intervention) and immediately post-intervention (within 30 minutes after the session)
  Change from baseline to immediate post-intervention, in the Attribution Questionnaire-27 (AQ-27) total score. Higher scores indicate greater explicit stigma toward individuals with schizophrenia.
  An immediate decrease in stigma scores on the AQ-27 in the intervention group compared to the control group is expected.
Implicit stigma - Immediate effect | Baseline (pre-intervention) and immediately post-intervention (within 30 minutes after the session)
  Change from baseline to immediate post-intervention, in implicit association between schizophrenia and violence, measured by the Implicit Association Test (IAT) score (higher absolute score indicates stronger implicit association). A greater immediate reduction in implicit associations linking schizophrenia with violence is expected in the intervention group compared to controls.
Attitudes toward individuals with schizophrenia - 1 month follow up | Baseline and 1 month follow-up
  Change from baseline to immediate post-intervention, in the Community Attitudes toward the Mentally Ill (CAMI) total score. Higher scores indicate more bad attitudes toward individuals with schizophrenia. An immediate decrease in stigma scores on the CAMI in the intervention group compared to the control group is expected.
Behaviors toward individuals with schizophrenia - 1 month follow up | Baseline and 1 month follow-up
  Change from baseline to immediate post-intervention, in the Reported and Intended Behavior Scale (RIBS) total score. Higher scores indicate more bad behaviors toward individuals with schizophrenia. An immediate decrease in stigma scores on the RIBS in the intervention group compared to the control group is expected.
Attitudes toward individuals with schizophrenia - immediate effect | Baseline (pre-intervention) and immediately post-intervention (within 30 minutes after the session)
  Change from baseline to immediate post-intervention, in the Community Attitudes toward the Mentally Ill (CAMI) total score. Higher scores indicate more bad attitudes toward individuals with schizophrenia. An immediate decrease in stigma scores on the CAMI in the intervention group compared to the control group is expected
Behaviors toward individuals with schizophrenia - immediate effect | Baseline (pre-intervention) and immediately post-intervention (within 30 minutes after the session)
  Change from baseline to immediate post-intervention, in the Reported and Intended Behavior Scale (RIBS) total score. Higher scores indicate more bad behaviors toward individuals with schizophrenia. An immediate decrease in stigma scores on the RIBS in the intervention group compared to the control group is expected.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Recherche Clinique (URC), Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared upon reasonable request for non-commercial research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available starting 6 months after publication for 36 months.
Access Criteria: Requests reviewed by the study team; data use agreement and IRB/ethics approval required.